CLINICAL TRIAL: NCT07209254
Title: Randomized Controlled Trial of Two Mobile Health Strategies to Manage Postpartum Hypertension
Acronym: SMART BP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Lewey, MD, MPH (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jennifer Lewey, MD, MPH, Assistant Professor of Medicine (Cardiovascular Medicine), University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 858860
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypertension, Pregnancy Induced
Keywords: Postpartum Hypertension; Blood pressure management; Preeclampsia; Hypertension, pregnancy induced
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-touch blood pressure management (Experimental)
  Interventions: Other: High-touch blood pressure management
- Low-touch blood pressure management (Experimental)
  Interventions: Other: Low-touch blood pressure management

INTERVENTIONS:
Other: High-touch blood pressure management — Twelve weeks of text-based home blood pressure monitoring with BP self-management and team-based care
  Arms: High-touch blood pressure management
Other: Low-touch blood pressure management — 10 days of text-based home blood pressure monitoring
  Arms: Low-touch blood pressure management

SUMMARY:
A multicenter randomized trial that will compare the effectiveness of two postpartum blood pressure (BP) management strategies in improving blood pressure and cardiac function and increasing patient engagement and feeling of control over one's health

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Delivery within 14 days
* Diagnosis of preeclampsia or gestational hypertension with or without severe features during pregnancy or within 14 days postpartum
* Initiation of blood pressure medication prior to hospital discharge and up to 14 days postpartum
* English or Spanish speaking (able to read/understand consent and instructions)
* Has phone texting capabilities

Exclusion Criteria:

* Diagnosis of chronic hypertension prior to delivery (would therefore include super imposed preeclampsia)
* Pre-existing cardiovascular disease (including prior myocardial infarction, stroke, heart failure with reduced ejection fraction, ventricular tachycardia, prior cardiac arrest, pacemaker, severe valvular heart disease, or prior cardiac surgery)
* Chronic kidney disease (stage 3 or higher)
* Using ≥3 BP medications at time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Mean diastolic blood pressure (DBP) | 12 months postpartum
  Assessed by 24-hour ambulatory blood pressure monitor (ABPM)

SECONDARY OUTCOMES:
Blood pressure outcome: Mean systolic blood pressure (SBP) | 12 months postpartum
  Assessed by 24-hour ambulatory blood pressure monitor (ABPM)
Blood pressure outcome: Mean nocturnal DBP | 12 months postpartum
  Assessed by ABPM
Blood pressure outcome: Mean nocturnal SBP | 12 months postpartum
  Assessed by ABPM
Blood pressure outcome: Mean DBP | 12 months postpartum
  Assessed by home blood pressure monitor and office measurement
Chronic Hypertension | 12 months postpartum
  Defined as 24-hour mean systolic blood pressure greater than or equal to 12mmHg, mean diastolic blood pressure greater than or equal to 75mmHg as assessed by ABPM or taking BP medication
Echocardiogram Outcomes | 12 months postpartum
  Patients will all undergo a routine transthoracic echocardiogram. Measurements include: Left ventricle (LV) mass index, Relative wall thickness, mean E/e' ratio, left atrial (LA) volume index, global longitudinal strain.
Patient Reported Outcome - Patient Activation Measure | Post-randomization to 1 year postpartum
  Patient Activation Measure (PAM) is a 10 survey that assesses an individual's knowledge, skills and confidence integral to managing one's own health and healthcare. Scored on a scale from 0-100 that correlates to one of four levels of patient activation. PAM Levels 1 and 2 indicate lower patient activation, while PAM Levels 3 and 4 indicate higher patient activation.
  Survey will be completed at 3 timepoints: at randomization, 6-10 weeks postpartum, and 12 months postpartum
Patient Reported Outcome - Perceived Stress | Post-randomization to 1 year postpartum
  Scores from the validated Perceived Stress Scale (PSS-10) will be calculated using standard scoring criteria for each of the 10 items. Higher scores are correlated with more perceived stress.
  Survey to be completed at randomization, at 6-10 weeks postpartum, and at 1 year postpartum.
Patient Reported Outcome - Self-Efficacy | Post randomization to 1 year postpartum
  New General Self-Efficacy Scale is an 8-item measure that assesses how much people believe they can achieve their goals, despite difficulties. Using a 5-point rating scale where 1=strongly disagree and 5=strongly agree, scores are calculated by taking the average of their ratings. Survey to be completed at randomization, at 6-10 weeks postpartum, and at 1 year postpartum.
Implementation Outcome: Acceptability of Intervention | From 6 weeks postpartum through 1 year postpartum
  Patients will be asked questions to assess the acceptability of the intervention. The questions will be scored on a Likert response scales from 1 to 5. Higher scores represent higher acceptability. Asked at two time points, 6 weeks and 12 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lewey, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - New York University, New York, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes